Statistical Analysis Plan version 2 H8H-MC-LAHU

A Randomized, Double-Blind, Four-Period, Crossover Study to Evaluate the Cardiovascular

Effect of Single Oral Doses of Lasmiditan when Coadministered with Single Oral Doses of

Sumatriptan in Healthy Subjects

NCT03310411

Approval Date: 22-Nov-2017

# STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Four-Period, Crossover Study to Evaluate the Cardiovascular Effect of Single Oral Doses of Lasmiditan when Coadministered with Single Oral Doses of Sumatriptan in Healthy Subjects

> Statistical Analysis Plan Status: Final v2 Statistical Analysis Plan Date: 02-Nov-2017

Study Drug: LY573144 (Lasmiditan)

Sponsor Reference: H8H-MC-LAHU Covance CRU Study: 1000071-8370358

Clinical Phase I

Approval Date: 22-Nov-2017 GMT

Final v2, 02 Nov 2017 

# 1. TABLE OF CONTENTS

| 1. | TAB | LE OF CONTENTS | 2 |
|----|-------|---------------------------------------------------|----------|
| 2. | | REVIATIONS | |
| 3. | INTR | ODUCTION | <i>6</i> |
| 4. | STUI | DY OBJECTIVES | <i>6</i> |
| | | Primary Objective | |
| | | Secondary Objectives | |
| | 4.3 E | Exploratory Objective | <i>6</i> |
| 5. | STUI | DY DESIGN | 7 |
| 6. | | ATMENTS | |
| 7. | SAM | PLE SIZE JUSTIFICATION | 8 |
| 8. | DEFI | NITION OF ANALYSIS POPULATIONS | 8 |
| 9. | STAT | FISTICAL METHODOLOGY | 8 |
| | 9.1 | General | 8 |
| | 9.2 I | Demographics and Subject Disposition | 9 |
| | 9.3 P | Pharmacokinetic Assessment | 9 |
| | 9.3. | 1 Pharmacokinetic Analysis | 9 |
| | 9.3. | 2 Pharmacokinetic Statistical Methodology | 13 |
| | 9.4 | Cardiovascular Assessment | 14 |
| | 9.4. | 1 Cardiovascular Analyses | 14 |
| | 9.4. | 2 Cardiovascular Statistical Methodology | 14 |
| | 9.5 S | afety and Tolerability Assessments | 15 |
| | 9.5. | 1 Adverse events | 15 |
| | 9.5. | 2 Concomitant medication | 16 |
| | 9.5. | 3 Clinical laboratory parameters | 16 |
| | 9.5. | 4 Hepatic Monitoring | 16 |
| | 9.5. | 5 Vital signs | 16 |
| | 9.5. | 6 Electrocardiogram (ECG) | 17 |
| | 9.5. | 7 Other assessments | 17 |
| | 9.5 | 8 Safety and Tolerability Statistical Methodology | 17 |

# CONFIDENTIAL Sponsor Reference H8H-MC-LAHU

| 9.6 Biomarker Analyses | 17 |
|-----------------------------------------------------|------------|
| 10. INTERIM ANALYSES | 17 |
| 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL | ANALYSES17 |
| 12. REFERENCES | 17 |
| 13. DATA PRESENTATION | 17 |
| 13.1 Derived Parameters | 17 |
| 13.2 Missing Data | 17 |
| 13.3 Insufficient Data for Presentation | |

Final v2, 02 Nov 2017 

## 2. ABBREVIATIONS

Abbreviations pertain to the Statistical Analysis Plan (SAP) only (not the tables, figures and listings [TFLs]).

ABP Ambulatory blood pressure

ABPM Ambulatory blood pressure monitoring

AE Adverse event

ALP Alkaline phosphatase

ALT Alanine aminotransferase

AUC Area under the concentration versus time curve

 $AUC(0-\infty)$  Area under the concentration versus time

 $AUC(0-t_{last})$  Area under the concentration versus time curve from time zero to

time t, where t is the last time point with a measurable concentration

%AUC(tlast- $\infty$ ) Percentage of AUC(0- $\infty$ ) extrapolated

BQL Below lower limit of quantitation

CI Confidence interval

C<sub>max</sub> Maximum observed drug concentration

CL/F Apparent total body clearance of drug calculated after extra-vascular

administration

CRF Case Report Form

CSR Clinical Study Report
CRU Clinical Research Unit
CV Coefficient of variation
DBP Diastolic blood pressure

EC Early Clinical

ECG Electrocardiogram

e.g. For example (Latin: *exempli gratia*)

ICH International Council on Harmonisation

LLOQ Lower limit of quantification

LS Least square

MAP Mean arterial pressure

MedDRA Medical Dictionary for Regulatory Activities

Final v2, 02 Nov 2017 

| MRE | Magnetic resonance elastography |
|---|---|
| PK | Pharmacokinetic |
| PR | Pulse rate |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SOP | Standard Operating Procedure |
| TBL | Total bilirubin |
| TFLs | Tables, Figures, and Listings |
| $t_{1/2}$ | Half-life associated with the terminal rate constant $(\lambda_z)$ in non-compartmental analysis |
| $t_{max}$ | Time of maximum observed drug concentration |
| ULN | Upper limit of normal |
| Vss/F | Apparent volume of distribution at steady state after extra-vascular administration |
| V <sub>z</sub> /F | Apparent volume of distribution during the terminal phase after extra-vascular administration |
| WHO | World Health Organization |

Final v2, 02 Nov 2017 

#### 3. INTRODUCTION

This SAP has been developed after review of the Clinical Study Protocol (final version dated 17 August 2017) and Protocol Amendment (c) (final version dated 20 October 2017).

This SAP describes the planned analysis of the safety, tolerability and pharmacokinetic (PK) data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical and PK analyses of data. In general, the analyses are based on information from the protocol, unless they have been modified by agreement between Eli Lilly and Company and Covance Early Clinical (EC) Biometrics. A limited amount of information concerning this study (e.g., objectives, study design) is given to help the reader's interpretation. This SAP must be signed off prior to first subject administration for this study. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified in the CSR. Any substantial deviations from this SAP will be agreed upon between Eli Lilly and Company and Covance EC Biometrics and identified in the CSR. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Council on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

## 4. STUDY OBJECTIVES

## 4.1 Primary Objective

• To compare and contrast the cardiovascular effects of lasmiditan 200 mg and sumatriptan 100 mg administered together to the cardiovascular effects of single doses of either drug administered alone.

# 4.2 Secondary Objectives

- To evaluate the PK of lasmiditan 200 mg and sumatriptan 100 mg administered either alone or together.
- To evaluate the safety and tolerability of lasmiditan 200 mg and sumatriptan 100 mg.

# 4.3 Exploratory Objective

- To evaluate the effect of lasmiditan on renal function biomarkers in serum and urine.
- To evaluate the PK of lasmiditan metabolites alone and in combination with sumatriptan in healthy subjects.

Final v2, 02 Nov 2017 

#### 5. STUDY DESIGN

This is a randomized, double-blind, crossover study with 4 study periods in healthy subjects. All subjects will participate in 4 treatment periods. The treatments are as follows:

- Treatment A: lasmiditan 200 mg + sumatriptan 100 mg
- Treatment B: lasmiditan 200 mg + placebo
- Treatment C: sumatriptan 100 mg + placebo
- Treatment D: placebo + placebo

Each subject will be randomized to one of 4 treatment sequences in a William's square design as outlined in Table 1.

**Table 1. Sequences in Study LAHU** 

| Sequence | Period 1 | Period 2 | Period 3 | Period 4 |
|----------|---------------|---------------|---------------|---------------|
| 1 | Lasmiditan + | Lasmiditan + | Sumatriptan + | Placebo + |
| | sumatriptan | placebo | placebo | placebo |
| 2 | Lasmiditan + | Sumatriptan + | Placebo + | Lasmiditan + |
| | placebo | placebo | placebo | sumatriptan |
| 3 | Sumatriptan + | | Lasmiditan + | Lasmiditan + |
| | placebo | placebo | sumatriptan | placebo |
| 4 | 4 Placebo + | | Lasmiditan + | Sumatriptan + |
| | placebo | sumatriptan | placebo | placebo |

# **Screening Period:**

All subjects will participate in a screening visit up to 28 days prior to Period 1 study drug dosing.

## **Treatment Periods:**

All subjects will participate in 4 treatment periods. Subjects will be randomized to one of 4 treatment sequences. They will be admitted to the clinical research unit (CRU) the day prior to dosing (Day -1) in Period 1, and will be dosed on Day 1 of each treatment period according to their assigned treatment sequence (Table 1). Subjects will be discharged from the CRU on Day 3 of Period 4 following the collection of all ambulatory blood pressure (ABP) measurements and PK blood samples.

There will be a washout of at least 4 days between each dosing day.

All subjects will be discharged from the study at least 5 days after discharge from Period 4.

Final v2, 02 Nov 2017 

#### 6. TREATMENTS

The following is a list of the study treatment abbreviations that will be used in the TFLs.

| Study Treatment Name | Treatment order in TFL |
|----------------------------------------|------------------------|
| Placebo | 1 |
| 200 mg lasmiditan + 100 mg sumatriptan | 2 |
| 200 mg lasmiditan + placebo | 3 |
| 100 mg sumatriptan + placebo | 4 |

#### 7. SAMPLE SIZE JUSTIFICATION

Up to 40 subjects may be enrolled to ensure 30 subjects complete the study. Assuming standard deviation for the change, within-subject, in systolic blood pressure (SBP) of 12.7 mmHg (based on results from study CCI with the power of the study of the st

#### 8. DEFINITION OF ANALYSIS POPULATIONS

The "Safety" population will consist of all enrolled subjects, whether or not they completed all protocol requirements.

The "Pharmacokinetic" population will consist of all subjects who received at least one dose of lasmiditan or sumatriptan and have evaluable PK data. Subjects may be excluded from the PK summary statistics and statistical analysis if a subject has an adverse event (AE) of vomiting that occurs at or before 2 times median time of maximum observed drug concentration (t<sub>max</sub>).

All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when subjects are assigned to analysis populations.

#### 9. STATISTICAL METHODOLOGY

## 9.1 General

Data listings will be provided for all data that is databased. Summary statistics and statistical analysis will only be presented for data where detailed in this SAP. For continuous data, summary statistics will include the arithmetic mean, arithmetic standard deviation (SD), median, min, max and N; for log-normal data (e.g. the PK parameters: area under the concentration versus time curve [AUCs] and maximum observed drug concentration [C<sub>max</sub>]) the geometric mean and geometric coefficient of variation (CV%) will also be presented. For categorical data, frequency count and percentages will be presented. Data listings will be provided for all subjects up to the point of withdrawal, with any subjects excluded from the relevant population

Final v2, 02 Nov 2017 

highlighted. Summary statistics and statistical analyses will generally only be performed for subjects included in the relevant analysis population. For the calculation of summary statistics and statistical analysis, unrounded data will be used.

Mean change from baseline is the mean of all individual subjects' change from baseline values. Each individual change from baseline will be calculated by subtracting the individual subject's baseline value from the value at the timepoint. The individual subject's change from baseline values will be used to calculate the mean change from baseline using a SAS procedure such as Proc Univariate.

Data analysis will be performed using SAS® Version 9.3 or greater.

# 9.2 Demographics and Subject Disposition

Subject disposition will be listed. The demographic variables age, sex, race, ethnicity, country of enrolment, site ID, body weight, height and body mass index will be summarized and listed.

## 9.3 Pharmacokinetic Assessment

# 9.3.1 Pharmacokinetic Analysis

PK parameter estimates will be determined using non-compartmental procedures in validated software program (Phoenix WinNonlin Version 6.4 or later).

Plasma concentrations of lasmiditan (LY573144), its metabolites, and sumatriptan will be used to determine the following PK parameters, when possible:

Final v2, 02 Nov 2017 

| Parameter | Units | Definition |
|---|---|---|
| C <sub>max</sub> | ng/mL | maximum observed drug concentration |
| t <sub>max</sub> | h | time of maximum observed drug concentration |
| AUC(0-∞) | ng.h/mL | area under the concentration versus time curve from time zero to infinity |
| AUC(0-t <sub>last</sub> ) | ng.h/mL | area under the concentration versus time curve from time zero to<br>time t, where t is the last time point with a measurable<br>concentration |
| $%AUC(t_{last}-\infty)$ | % | percentage of AUC(0-∞) extrapolated |
| $\mathbf{t}_{_{1\!/_{\!2}}}$ | h | half-life associated with the terminal rate constant $(\lambda_z)$ in non-compartmental analysis |
| CL/F | L/h | apparent total body clearance of drug calculated after extra-vascular administration (LY573144 and sumatriptan only) |
| $V_z/F$ | L | apparent volume of distribution during the terminal phase after extra-vascular administration (LY573144 and sumatriptan only) |
| $V_{ss}/F$ | L | apparent volume of distribution at steady state after extra-vascular administration (LY573144 and sumatriptan only) |
| MR | | Metabolic ratio <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup> = no molar correction will be applied since the metabolites are very similar in molecular weight and within 5% of the molecular weight for lasmiditan.

Additional PK parameters may be calculated, as appropriate. The software and version used for the final analyses will be specified in the CSR. Any exceptions or special handling of data will be clearly documented within the final study report.

Formatting of tables, figures and abbreviations will follow the Eli Lilly Global PK/PD/TS Tool: NON-COMPARTMENTAL PHARMACOKINETIC STYLE GUIDE. The version of the tool effective at the time of PK analysis will be followed.

## **General PK Parameter Rules**

- Actual sampling times will be used in the final analyses of individual PK parameters, except for non-bolus pre-dose sampling times which will be set to zero.
- $C_{max}$  and  $t_{max}$  will be reported from observed values. If  $C_{max}$  occurs at more than one time point,  $t_{max}$  will be assigned to the first occurrence of  $C_{max}$ .
- AUC parameters will be calculated using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule). The linear trapezoidal method will be applied up to t<sub>max</sub> and then the logarithmic trapezoidal method will be used after t<sub>max</sub>. The minimum requirement for the calculation of AUC will be the inclusion of at least three consecutive plasma concentrations above the lower limit of quantification (LLOQ), with at least one of these concentrations following C<sub>max</sub>. AUC(0-∞) values where the

Final v2, 02 Nov 2017 

percentage of the total area extrapolated is more than 20% will be flagged. Any  $AUC(0-\infty)$  value excluded from summary statistics will be noted in the footnote of the summary table.

- Half-life (t<sub>1/2</sub>) will be calculated, when appropriate, based on the apparent terminal log-linear portion of the concentration-time curve. The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in plasma concentrations. Half-life will only be calculated when a reliable estimate for this parameter can be obtained comprising of at least 3 data points. If t<sub>1/2</sub> is estimated over a time window of less than 2 half-lives, the values will be flagged in the data listings. Any t<sub>1/2</sub> value excluded from summary statistics will be documented in the footnote of the summary table.
- A uniform weighting scheme will be used in the regression analysis of the terminal loglinear portion of the concentration-time curve.
- The parameters based on predicted C<sub>last</sub> will be reported.

## **Individual PK Parameter Rules**

- Only quantifiable concentrations will be used to calculate PK parameters with the exception of special handling of certain concentrations reported below the lower limit of quantitation (BQL). Plasma concentrations reported as BQL will be set to a value of zero when all of the following conditions are met:
  - The compound is non-endogenous.
  - The samples are from the initial dose period for a subject or from a subsequent dose period following a suitable wash-out period.
  - o The time points occur before the first quantifiable concentration.
- All other BQL concentrations that do not meet the above criteria will be set to missing.
- Also, where two or more consecutive concentrations are BQL towards the end of a profile, the profile will be deemed to have terminated and therefore any further quantifiable concentrations will be set to missing for the calculation of the PK parameters unless it is considered to be a true characteristic of the profile of the drug.

## **Individual Concentration vs. Time Profiles**

- Individual concentrations will be plotted utilizing actual sampling times.
- The terminal point selections will be indicated on a semi-logarithmic plot.

Final v2, 02 Nov 2017 

## **Average Concentration vs. Time Profiles**

- The average concentration profiles will be graphed using scheduled (nominal) sampling times.
- The average concentration profiles will be graphed using arithmetic average concentrations.
- The pre-dose average concentration for single-dose data from non-endogenous compounds will be set to zero.
- Concentrations at a sampling time exceeding the sampling time window specified in the protocol, or  $\pm$  10%, will be excluded from the average concentration profiles.
- Concentrations excluded from the mean calculation will be documented in the final study report.
- A concentration average will be plotted for a given sampling time only if 2/3 of the individual data at the time point have quantifiable measurements that are within the sampling time window specified in the protocol or ± 10%. An average concentration estimated with less than 2/3 but more than 3 data points may be displayed on the mean concentration plot if determined to be appropriate and will be documented within the final study report.

# **Treatment of Outliers during Pharmacokinetic Analysis**

Application of this procedure to all PK analyses is not a requirement. Rather, this procedure provides justification for exclusion of data when scientifically appropriate. This procedure describes the methodology for identifying an individual value as an outlier for potential exclusion, but does not require that the value be excluded from analysis. The following methodology will not be used to exclude complete profiles from analysis.

## Data within an Individual Profile

A value within an individual profile may be excluded from analysis if any of the following criteria are met:

- For PK profiles during single dosing of non-endogenous compounds, the concentration in a pre-dose sample is quantifiable.
- For any questionable datum that does not satisfy the above criteria, the profile will be evaluated and results reported with and without the suspected datum.

## Data between Individual Profiles

1. If n<6, then the dataset is too small to conduct a reliable range test. Data will be analyzed with and without the atypical value, and both sets of results will be reported.

Final v2, 02 Nov 2017 

- 2. If n≥6, then an objective outlier test will be used to compare the atypical value to other values included in that calculation:
  - a. Transform all values in the calculation to the logarithmic domain.
  - b. Find the most extreme value from the arithmetic mean of the log transformed values and exclude that value from the dataset.
  - c. Calculate the lower and upper bounds of the range defined by the arithmetic mean  $\pm 3*SD$  of the remaining log-transformed values.
  - d. If the extreme value is within the range of arithmetic mean  $\pm 3*SD$ , then it is not an outlier and will be retained in the dataset.
  - e. If the extreme value is outside the range of arithmetic mean  $\pm 3*SD$ , then it is an outlier and will be excluded from analysis.

If the remaining dataset contains another atypical datum suspected to be an outlier and  $n \ge 6$  following the exclusion, then repeat step 2 above. This evaluation may be repeated as many times as necessary, excluding only one suspected outlier in each iteration, until all data remaining in the dataset fall within the range of arithmetic mean  $\pm 3*SD$  of the log-transformed values.

# Reporting of Excluded Values

Individual values excluded as outliers will be documented in the final report. Approval of the final report will connote approval of the exclusion.

# 9.3.2 Pharmacokinetic Statistical Methodology

PK parameter estimates will be evaluated to determine the impact of a single oral dose of sumatriptan 100 mg on the PK of lasmiditan and its metabolites. Log-transformed  $C_{max}$ ,  $AUC(0-\infty)$ , and  $AUC(0-t_{last})$  will be evaluated using a linear effects model with fixed effects for treatment, period (1, 2, 3, or 4) and treatment sequence, and a random effect for subject. From this model, the 90% CI of the ratio of geometric means from Treatment A (lasmiditan + sumatriptan) will be determined and presented versus those of Treatment B (lasmiditan + placebo).

An example of the SAS code that will be used is as follows:

```
proc mixed data=xxx;
  by analyte;
  class trtmnt period seq subject;
  model l_pk = trtmnt period seq / alpha=0.1;
  random subject;
  lsmeans trtmnt / pdiff;
run;
```

where 1 pk is the log-transformed (base e) PK parameter.

Final v2, 02 Nov 2017 

The  $t_{max}$  will be analyzed using a Wilcoxon signed rank test. Estimates of the median difference based on the observed medians, 90% CIs, and the p-values from the Wilcoxon test will be calculated.

The same model will be independently used to assess the impact of a single oral dose of lasmiditan 200 mg on the PK of single oral dose of sumatriptan 100 mg.

Additional analyses may be performed, as warranted.

## 9.4 Cardiovascular Assessment

## 9.4.1 Cardiovascular Analyses

The primary parameters for the cardiovascular analyses will be peak hourly mean values of SBP, diastolic blood pressure (DBP), and mean arterial pressure (MAP), and nadir hourly mean values for pulse rate (PR), and will be determined by ambulatory blood pressure monitoring (ABPM). These data will be listed and summarized by treatment.

Mean hourly SBP, DBP, MAP, and PR values will be calculated, summarized by treatment, and plotted, together with changes from baseline. Baseline value will be defined as the mean value during the 2 hours pre-dose for each period.

Finally, descriptive statistics will be used to summarize the mean values of SBP, DBP, MAP, and PR parameters over the intervals 0-4 h, 4-8h, 8-12 h, and 12-24 h.

## 9.4.2 Cardiovascular Statistical Methodology

## **Primary analysis**

Changes from baseline in peak hourly mean values of cardiovascular parameters SBP, DBP, and MAP, and nadir hourly mean values of PR will be analysed to determine the impact of a single dose of sumatriptan 100 mg on the peak/nadir hourly mean values of the cardiovascular parameters of lasmiditan. A linear mixed-effects model with baseline as a covariate, fixed effects for treatment, period (1, 2, 3, or 4), and treatment sequence, and a random effect for subject will be used. Least squares (LS) means and treatment differences ([lasmiditan + sumatriptan] - [lasmiditan + placebo]) will be calculated and presented with the corresponding CIs.

Primary cardiovascular parameters may be log-transformed prior to the statistical analysis if a review of the data indicates that the assumption of normality is violated.

The same model will be used to assess the impact of a single dose of lasmiditan 200 mg on the peak/nadir hourly mean values of the cardiovascular parameters of sumatriptan.

Final v2, 02 Nov 2017 

An example of the SAS code that will be used is as follows:

```
proc mixed data=xxx;
    class trtmnt period seq subject;
    model primcard = base trtmnt period seq / alpha=0.1 cl ddfm=kr;
    random subject;
    lsmeans trtmnt / alpha=0.1 cl pdiff;
run;
```

where 'primard' is the change from baseline in the peak/nadir hourly mean values of the primary cardiovascular parameters SBP, DBP, MAP/PR respectively.

# Repeated measures analysis:

Changes from baseline in cardiovascular parameters will be evaluated to determine the impact of a single oral dose of sumatriptan 100 mg on the cardiovascular parameters of single oral dose of lasmiditan 200 mg.

A repeated measures linear mixed-effects model with baseline as a covariate, fixed effects for time point, treatment, period (1, 2, 3, or 4), treatment sequence, and the treatment by time point interaction, and a random effect for subject will be used. LS means and treatment differences ([lasmiditan + sumatriptan] – [lasmiditan + placebo]) will be calculated and presented with the corresponding 90% CIs.

An example of the SAS code that will be used is as follows:

```
proc mixed data=xxx;
    class trtmnt subject time period seq;
    model cardio = base time trtmnt period seq trtmnt*time / alpha=0.1 cl ddfm=kr;
    repeated time / type=un subject=subject;
    random subject;
    lsmeans trtmnt*time / alpha=0.1 cl pdiff;
run;
```

where 'cardio' is the change from baseline in the cardiovascular parameter.

Cardiovascular parameters may be log-transformed prior to the statistical analysis if a review of the data indicates that the assumption of normality is violated.

The same model will be used to assess the impact of a single dose of lasmiditan 200 mg on the cardiovascular parameters of sumatriptan.

# 9.5 Safety and Tolerability Assessments

## 9.5.1 Adverse events

Where changes in severity are recorded in the Case Report Form (CRF), each separate severity of the AE will be reported in the listings, only the most severe will be used in the summary tables. A pre-existing condition is defined as an AE that starts before the subject has provided written informed consent and is ongoing at consent. A non-treatment emergent AE is defined as an AE which starts after informed consent but prior to dosing. A treatment-emergent AE is

Final v2, 02 Nov 2017 

defined as an AE which occurs postdose or which is present prior to dosing and becomes more severe postdose.

All AEs will be listed. Treatment-emergent AEs will be summarized by treatment, severity and relationship to the study drug. The frequency (the number of AEs, the number of subjects experiencing an AE and the percentage of subjects experiencing an AE) of treatment-emergent AEs will be summarized by treatment, Medical Dictionary for Regulatory Activities (MedDRA) version 20.0 system organ class and preferred term. The summary and frequency AE tables will be presented for all causalities and those considered related to the study drug. Any serious AEs will be tabulated.

## 9.5.2 Concomitant medication

Concomitant medication will be coded using the WHO drug dictionary (Version March 2017 Enhanced Dictionary B2 Format). Concomitant medication will be listed.

## 9.5.3 Clinical laboratory parameters

All clinical chemistry, hematology and urinalysis data will be listed. Additionally clinical chemistry, hematology and urinalysis data outside the reference ranges will be listed.

Values for any clinical chemistry, hematology and urinalysis values outside the reference ranges will be flagged on the individual subject data listings.

# 9.5.4 Hepatic Monitoring

If a subject experiences elevated alanine aminotransferase (ALT)  $\ge 3 \times$  upper limit of normal (ULN), alkaline phosphatase (ALP)  $\ge 2 \times$  ULN, or elevated total bilirubin (TBL)  $\ge 2 \times$  ULN, liver tests will be performed to confirm the abnormality.

The subjects' liver disease history and associated person liver disease history data will be listed. Any concomitant medication of acetaminophen/paracetamol will be listed. Results from any hepatic monitoring procedures, such as a magnetic resonance elastography (MRE) scan, and a biopsy assessment will be listed, if performed.

Hepatic risk factor assessment data will be listed. Liver related signs and symptoms data will be summarized by treatment and listed. Alcohol and recreational drug use data will also be listed.

All hepatic chemistry, hematology, coagulation, and serology data will be listed. Values outside the reference ranges will be flagged on the individual subject data listings.

# 9.5.5 Vital signs

Supine vital signs data will be summarized by treatment together with changes from baseline, where baseline is defined as Day 1 predose. Furthermore, values for individual subjects will be listed.

Final v2, 02 Nov 2017 

# 9.5.6 Electrocardiogram (ECG)

For each subject, ECGs will be performed for safety purposes only, and will not be reported.

#### 9.5.7 Other assessments

All other safety assessments not detailed in this section will be listed but not summarized or statistically analyzed.

# 9.5.8 Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

# 9.6 Biomarker Analyses

Exploratory biomarkers such as creatinine clearance and renal biomarkers, including, but not limited to, creatinine and cystatin C levels, will be summarized by treatment and listed.

## 10. INTERIM ANALYSES

No interim statistical analyses are planned.

## 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES

There were no changes from the protocol specified statistical analyses.

## 12. REFERENCES

- 1. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.
- 2. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.

## 13. DATA PRESENTATION

## 13.1 Derived Parameters

Individual derived parameters (e.g. PK parameters) and appropriate summary statistics will be reported to three significant figures. Observed concentration data, e.g.  $C_{max}$ , should be reported as received. Observed time data, e.g.  $t_{max}$ , should be reported as received. N and percentage values should be reported as whole numbers. Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

# 13.2 Missing Data

Missing data will not be displayed in listings.

Final v2, 02 Nov 2017 

# 13.3 Insufficient Data for Presentation

Some of the TFLs may not have sufficient numbers of subjects or data for presentation. If this occurs, the blank TFL shell will be presented with a message printed in the centre of the table, such as, "No serious adverse events occurred for this study."

Final v2, 02 Nov 2017 

## Leo Document ID = 0aca3db4-3fe8-4725-b16a-552cce8ea5e1

Approver: PPD

Approval Date & Time: 13-Nov-2017 10:31:51 GMT Signature meaning: Approved

Approver: PPD

Approval Date & Time: 13-Nov-2017 13:19:29 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 13-Nov-2017 13:36:27 GMT

Signature meaning: Approved

Approver: PPD
Approval Date & Time: 22-Nov-2017 13:20:12 GMT
Signature meaning: Approved